CLINICAL TRIAL: NCT06615271
Title: Pressure Injuries in the Operating Room and Their Perioperative Incidence in Patients Undergoing Neurosurgery.
Acronym: UPS
Status: Recruiting | Type: Observational
Sponsor: Instituto de Investigación Marqués de Valdecilla (Other)
Responsible Party: Sponsor
Other Study IDs: UPS
Record Dates: First submitted 2023-10-24; First posted 2024-09-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: PRESSURE INJURIES
Keywords: injuries; surgical; neurosurgery; prevention; nurse; clinical practice
MeSH Terms: conditions — Pressure Ulcer; Wounds and Injuries | interventions — Neurosurgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who have undergone neurosurgery form more than 3 hours.: The ones who perform the selection criteria determined for this study will be chosen consecutively, and a follow-up will be carried out from the immediate preoperative moment until 72 hours once the surgery has finished.
  Interventions: Procedure: Neurosurgery

INTERVENTIONS:
Procedure: Neurosurgery — Patients who have undergone neurosurgery form more than 3 hours.

SUMMARY:
This research project is a descriptive, longitudinal prospective observational study in the HUMV neurosurgery operating rooms. The patients included will be adults 18 years old or older, who will be scheduled for surgery by the Neurosurgery service. Those who meet the selection criteria determined for this study will be chosen consecutively and will be followed from the immediate preoperative moment until 72 hours after the end of the surgery. Data collection shall be carried out by direct observation and immersion in clinical records of patients who have signed the informed consent. The study will be carried out in 4 phases: immediate preoperative, intraoperative, immediate postoperative and late postoperative, recording the data using various measuring instruments, and a record sheet. Finally, the cumulative incidence of LPPs developed in the perioperative environment will be calculated and a statistical analysis will be performed.

DETAILED DESCRIPTION:
The surgical area represents a scenario to be taken into account in the prevention of pressure injuries (LPP), being an essential and priority aspect in these injuries, demonstrating that more than 95% of them are avoidable. The latest national incidence study conducted in 2019, shows an incidence figure of 14% in post-surgical units and resuscitation, approaching the US between 12% and 66% of incidence in surgical patients, being considered a sentinel event, considering a medical cost of more than $26.8 billion.

The project will be developed from June 2023 to May 2025. It has been approved by the Research Ethics Committee of Cantabria, and the start of the study is scheduled for October 2023. Afterwards, the analysis of the data and the interpretation of the results will be done, ending with a final article to be disseminated and disseminated in magazines, congresses or national and international talks.

Surgical patients present specific risk factors, leading to the appearance of LPP. Therefore, this study aims to obtain some initial data to create a clinical care guide and prevention protocols updated and specific for clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients who understand and sign the informed consent.
* Adult patients of both sexes who will undergo a schedule surgery of more than 3 hours, by the service of neurosurgery of the University Hospital Marqués of Valdecilla (HUMV), between 2023 and 2024.
* Patients positioned in prone, supine, lateral and beach chair/sitting.
* Surgeries susceptible to bladder catheterisation with body temperature measurement.
* Patients admitted into neurosurgery ward, the day before surgery.

Exclusion Criteria:

* Patients who do not sign informed consent.
* Patients with visible pressure injurie present before surgery.
* Patients with cognitive disorder or written and oral knowledge difficulty.
* Patients who reject the operation.
* Patients not operated due to lack of prior time.
* Patients who do not receive vasoactive drugs such as ephedrine, phenylephrine and noradrenaline.
* Patients whose postoperative period is performed in the ICU.
* Patients whose surgical intervention, despite the initial estimate of the surgical time, lasted less than 3 hours.
* Patients admitted >24 hours prior the surgery.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients over 18 years, women and men.
Sampling Method: Non-Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of pressure injuries in the neurosurgery, in surgical interventions lasting more than 3 hours. It will be measured by direct observation of the wound, from the time the patient enters the operating room until the next 72 hours thereafter. | 72 hours

SECONDARY OUTCOMES:
Locations of the pressure injuries concerning to the different types of positioning.It will be measured by direct observation of the wound, from the time the patient enters the operating room until the next 72 hours thereafter. | 72 hours
the risk factors that contribute to the appearance of pressure injurieS. It will be measured by direct observation of the wound, from the time the patient enters the operating room until the next 72 hours thereafter. | 72 hours

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Hospital universitario marques de valdecilla, Santander

IPD SHARING:
Plan to Share IPD: No